CLINICAL TRIAL: NCT06950970
Title: Assessing the Effectiveness of Tion-Emo Therapy and Technique as a New Treatment Option for Depression and Anxiety
Brief Title: Evaluating the Effectiveness of Tion-Emo Therapy and Technique (TET)
Acronym: TET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rafael Navia (Other)
Responsible Party: Sponsor-Investigator, Rafael Navia, Investigator, TET Institute for development of psychotherapy and artificial emotion
Organization: TET Institute for development of psychotherapy and artificial emotion (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: TET Institute
Record Dates: First submitted 2025-04-06; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Depressive and Anxiety Disorders
Keywords: Objects, Therapy, comparison; Depression, Anxiety
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Methods

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm: "Patients receiving the investigational TET therapy and technique ." (Experimental): The experimental group received the TET therapy and technique based on its theoretical framework between 10 and 12 sessions for one hour each.
  Interventions: Behavioral: Tion-Emo therapy and technique for depression and anxiety Improvement
- Treatment Arm: "Patients not receiving the investigational TET therapy." (No Intervention): The patients did not receive any treatment, only pre-test and post-test.

INTERVENTIONS:
Behavioral: Tion-Emo therapy and technique for depression and anxiety Improvement — From 10 a 12 sessions once a week and one hour each session , for a positive result and development it is necessary to practice the technique
  Arms: Treatment Arm: "Patients receiving the investigational TET therapy and technique ."

SUMMARY:
The goal of this clinical trial is to explore the new therapy Cion-Emo therapy (TET) and to see if this technique is effective for treating depression and anxiety. Does TET lower anxiety and depression as participants learn and use this therapy? Researchers will compare TET with a control group to see if TET works in treating depression and anxiety. There was a pre-test and a post-test for both groups, experimental and control, and questionnaires to evaluate the effectiveness of TET. There was also a question to evaluate the hypothesis of the existence of nucleon emotion. The experimental group received TET therapy and techniques on an average of 10 to 12 one-hour sessions per week. The control group visited the clinic three times: in the first week all participants were evaluated to ascertain whether they were suffering from anxiety and depression; the second time was for the pre-test; and the third time was for the post-test.

DETAILED DESCRIPTION:
The TION-EMO theory (TET) was developed in Finland approximately four decades ago with positive results in the public and private sectors. Positive results were also seen in Ecuador. The psychological system is divided into three regions: the first is a self-survival region to regulate all emotions connected with survival. For example, when a person wants to avoid getting contaminated with COVID-19, the survival region is activated in to avoid contracting the disease. Another clear example occurs when people see a tiger- the first thing they want to do is escape. This example of survival mechanism is good; however, the bad effect is that in many cases the self-survival emotions remain long after the incident has occurred, causing a negative effect on health. Depression and anxiety are mostly affected by the social region- the area connected with humans' relations with the people they meet. Finally, people have the intellectual region. The author discovered that when people imagine themselves feeling their own body, they automatically make direct contact with the self-survival region. In the case of self-survival anxiety, people can imagine the object which is causing anxiety. Lately, investigators have noticed that people do not need this self-survival object because it does not have any responsibility. TET therapy addresses this self-survival object through supervised guidance by trained therapists. All this guidance has a very special effect on people's moods. In the case of anxieties and depressions caused by the social region, people imagine the self-object, that is, the individual plus the social object that is causing the anxiety or depression plus the supporting words, which can only be understandable phrases agreed upon by the patient and taught by the therapist. This process takes three to four sessions to understand the logic of the therapy. Several authors consider human objects to be important in the development of emotions, as well as their cognitive components in the comparison of the two. The research will focus on demonstrating that people who use the CION-EMO technique can regulate the symptoms of anxiety and depression caused by conflict and stress. This research is highly desirable.

ELIGIBILITY:
Inclusion: Confirmed diagnosis of depressive disorder or anxiety disorder: Based on clinical interview according to DSM criteria

* Age between 18 and 75 years
* Baseline symptom severity
* BAI score ≥ 22 (indicating at least moderate anxiety)
* Ability to attend intervention sessions for 12 weeks as part of the study protocol
* Informed consent signed before enrollment
* Exclusion Criteria: Diagnosis of bipolar disorder, schizophrenia, or psychotic disorders, as these conditions may require different treatment approaches and could confound results.
* Substance abuse or dependency, evaluated in the screaning interview.
* Severe neurological impairment or cognitive disorder, that may limit participation and affect the study outcomes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2025-02-08 (Actual)

PRIMARY OUTCOMES:
Reduction of depressive symptoms | Assessments will be conducted at baseline and 12 weeks post-treatment (pre-test and post-test), including comparisons with a control group.
  Assessment of the severity of depressive symptoms using the Beck Depression Inventory II (BDI-II), a self-report questionnaire with 21 items, each scored from 0 to 3. The total score ranges from 0 to 63, with interpretive ranges defined as:
  0-13: Minimal depression 14-19: Mild depression 20-28: Moderate depression 29-63: Severe depression Unit of Measure: Total score on the BDI-II.
  All statistical analyses were performed in R (v4.3) using:
  * ordinal: for modeling with a mixed ordinal regression approach
  * emmeans: for post hoc comparisons
  * MuMIn: for model fit metrics
  * ggplot2: for graphical display of results
Improvement in anxiety symptoms | Assessments will be conducted at baseline and 12 weeks post-treatment (pre-test and post-test), including comparisons with a control group.
  Measured using the Beck Anxiety Inventory (BAI), a self-report questionnaire consisting of 21 questions. Each item is scored from 0 to 3, yielding a total score range of 0 to 63. The suggested cut-off points for anxiety levels are:
  0-21: Very low anxiety 22-35: Moderate anxiety 36 and above: Severe anxiety Unit of Measure: Total score on the BAI.
  All statistical analyses were performed in R (v4.3) using:
  * ordinal: for modeling with a mixed ordinal regression approach
  * em means: for post hoc comparisons
  * MuMIn: for model fit metrics
  * ggplot2: for graphical display of results

SECONDARY OUTCOMES:
Effectiveness of the TET (Tion-Emo) technique for the control of depression | Assessments conducted at baseline and 12 weeks post-treatment (pre-test and post-test), including comparisons with a control group.
  Measured using the Questionnaire: "Evaluating the Effectiveness of TET" developed by the principal investigator and reviewed by two psychologists. The questionnaire consists of 12 items, each rated on a Likert scale ranging from 0 (not at all) to 10 (completely). will be summarized as percentages for each response category and analyzed for trends.
Effectiveness of the TET (Tion-Emo) technique in regulating anxiety | Assessments conducted at baseline and 12 weeks post-treatment (pre-test and post-test), including comparisons with a control group
  Measured using the Questionnaire: "Evaluating the Effectiveness of TET", developed by the principal investigator and reviewed by two psychologists. The questionnaire consists of 12 items, each rated on a Likert scale ranging from 0 (not at all) to 10 (completely). will be summarized as percentages for each response category and analyzed for trends.
Belief in the hypothesis of the core of emotions, this includes evaluating agreement with the statement: "All social emotions stem from the core of emotion." | Assessments will be conducted at baseline and 12 weeks post-treatment (pre-test and post-test), including comparisons with a control group.
  Measured by: "The questionnaire to evaluate the effectiveness of TET". Answers to all questions were evaluated on a Likert scale ranging from 0 (not at all) to 10 (completely). Data will be summarized as percentages for each response category and analyzed for trends.
1. Ease of using the TET technique | 4. Assessments will be conducted at baseline and 12 weeks post-treatment (pre-test and post-test), including comparisons with a control group.
  Measured by: "The questionnaire to evaluate the effectiveness of TET". Answers to all questions, were evaluated on a Likert scale ranging from 0 (not at all) to 10 (completely). Data will be summarized as percentages for each response category and analyzed for trends.
2. Ease of learning the TET technique | Assessments will be conducted at baseline and 12 weeks post-treatment (pre-test and post-test), including comparisons with a control group.
  Measured by: "The questionnaire to evaluate the effectiveness of TET". Answers to all questions, were evaluated on a Likert scale ranging from 0 (not at all) to 10 (completely). Data will be summarized as percentages for each response category and analyzed for trends.
3. General helpfulness of the TET technique | Assessments will be conducted at baseline and 12 weeks post-treatment (pre-test and post-test), including comparisons with a control group
  Measured by: "The questionnaire to evaluate the effectiveness of TET". Answers to all questions, were evaluated on a Likert scale ranging from 0 (not at all) to 10 (completely). Data will be summarized as percentages for each response category and analyzed for trends.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Navia, Principal Investigator — No afiliado
Locations (1):
- TET institute for development of psychotherapy and artificial emotion, Portoviejo, Manabí, Ecuador

IPD SHARING:
Plan to Share IPD: Yes
All data without breaking anonymity
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Deadline: Data requests can be submitted starting nine months after the article's publication and will be available for up to 24 months. Extensions are considered on a case-by-case basis.
Access Criteria: Qualified researchers conducting independent scientific research may request access to clinical trial research information (CRI). This access will be provided upon review and approval of a research proposal and Statistical Analysis Plan (SAP) and the signing of a Data Sharing Agreement (DSA). For more information or to submit a request.
URL: https://tionemoorg.wordpress.com/wp-admin/site-editor.php?canvas=edit&p=/

REFERENCES:
- [Background] Salvatore S, Tschacher W, Gelo OC, Koch SC. Editorial: Dynamic systems theory and embodiment in psychotherapy research. A new look at process and outcome. Front Psychol. 2015 Jul 1;6:914. doi: 10.3389/fpsyg.2015.00914. eCollection 2015. No abstract available. PMID 26191023
- [Background] Gilbert DT, Giesler RB, Morris KA. When comparisons arise. J Pers Soc Psychol. 1995 Aug;69(2):227-36. doi: 10.1037//0022-3514.69.2.227. PMID 7643304
- [Background] Spurio MG. The new functional identity: a body that thinks, a mind that feels - Frontiers and unexplored territories of the "Body and Mind zone". Psychiatr Danub. 2016 Sep;28(Suppl-1):111-115. PMID 27663819
- See also: Related Info — https://tionemoorg.wordpress.com/wp-admin/site-editor.php?canvas=edit&p=/
- Available data/document: Informed Consent Form: tetinstitute.rn@gmail.com — https://tionemoorg.wordpress.com/wp-admin/site-editor.php?canvas=edit&p=/
- Available data/document: Statistical Analysis Plan: tetinstitute.rn@gmail.com — https://tionemoorg.wordpress.com/wp-admin/site-editor.php?canvas=edit&p=/